CLINICAL TRIAL: NCT01949779
Title: TransForm™ Occlusion Balloon Catheter Registry
Status: Completed | Type: Observational
Sponsor: Stryker Neurovascular (Industry)
Responsible Party: Sponsor
Other Study IDs: T4023
Record Dates: First submitted 2013-09-20; First posted 2013-09-25 (Estimated); Results first posted 2019-08-19 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-08

CONDITIONS: Intracranial Aneurysms
Keywords: Coil embolization; TransForm™ Occlusion Balloon Catheter; Registry; Neurointerventional procedures
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TransForm™ Occlusion Balloon Catheter: TransForm™ Occlusion Balloon Catheter
  Interventions: Device: TransForm™ Occlusion Balloon Catheter

INTERVENTIONS:
Device: TransForm™ Occlusion Balloon Catheter — TransForm™ Occlusion Balloon Catheter

SUMMARY:
The primary objective of this registry is to collect real world data on the safety and performance of the TransForm™ Occlusion Balloon Catheter when used in current neurointerventional procedures

DETAILED DESCRIPTION:
* This is a prospective, single-arm, non-randomized, multi-center, observational registry.
* The expected duration for study enrollment is approximately 6 months-1 year.
* Study participation for each subject will be completed upon removal of the guide catheter post-procedure.
* Up to 140 subjects will be enrolled at up to 15 study sites. A given site will be allowed to enroll a maximum of 20 subjects.
* Enrollment in the registry occurs after a signed Informed Consent Form has been obtained, and the index procedure starts.

ELIGIBILITY:
Inclusion Criteria:

1. Subject or legal representative is willing and has provided informed consent.
2. Subject is scheduled to undergo a neurointerventional procedure that may include the use of the occlusion balloon catheter.
3. Subject is over 18 years of age.

Exclusion Criteria:

1. Subject's anatomy precludes safe delivery of the TransForm Occlusion Balloon Catheter.
2. Subject's pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care/hospitals
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2013-12; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (6):
  - Desert Regional Medical Center, Palm Springs, California
  - Central Baptist Hospital, Lexington, Kentucky
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - West Virginia University, Morgantown, West Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Hospital Universitario Donostia, Donostia / San Sebastian, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment occurred over 13 months at 7 sites in the US and 1 site in Spain. Each site was allowed to enroll up to 20 consecutive subjects. The first subject was enrolled on 12 December 2013 and the enrollment was completed on 12 January 2015. A total of 81 subjects were enrolled.
Groups:
- TransForm OBC: TransForm Occlusion Balloon Catheter
Period: Overall Study
Arm/Group | TransForm OBC
Started | 81
Completed | 79
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | TransForm OBC
Number analyzed (Participants) | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.78 (14.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 25
Region of Enrollment [Number; unit: participants]
  United States | 66
  Spain | 15

OUTCOME MEASURES:

1. Primary Outcome: Catheters Visualized That Reached Intended Target
Description: The number of TransForm™ OBC catheters that reached the intended target location confirmed by angiography visualization.
Time Frame: intra-procedure
Population: The number of catheters exceeds the number of participants enrolled, as more than one catheter may have been used for each participant.
Measure: Mean (Standard Deviation); unit: Catheters
Units Other Than Participants: Catheters
Groups:
- TransForm™ OBC: TransForm™ Occlusion Balloon Catheter
Arm/Group | TransForm™ OBC
Number analyzed (Participants) | 81
Number analyzed (Catheters) | 83
Catheters | 1.59 (0.78)

2. Secondary Outcome: Angiographic Assessment on Catheter
Description: Visibility of TransForm™ OBC on angiography
Time Frame: intra-procedure
Measure: Mean (Standard Deviation); unit: Catheters
Units Other Than Participants: Catheters
Arm/Group | TransForm™ OBC
Number analyzed (Participants) | 81
Number analyzed (Catheters) | 83
Catheters | 1.78 (0.84)

3. Secondary Outcome: Procedural Technical Success
Description: Ability of TransForm™ OBC to Perform as Intended
Time Frame: post-procedure
Measure: Number; unit: Catheters
Arm/Group | TransForm™ OBC
Number analyzed (Participants) | 81
Catheters | 83

ADVERSE EVENTS:
Arm/Group | TransForm OBC
Serious Adverse Events (participants affected / at risk) | 3/81
Other Adverse Events (participants affected / at risk) | 2/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TransForm OBC (N=81)
Thromboembolic event (Injury, poisoning and procedural complications) | 2
Vessel rupture/perforation (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TransForm OBC (N=81)
Thrombus formation (Surgical and medical procedures) | 1
Thrombus formation (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less